CLINICAL TRIAL: NCT00857090
Title: Double-Blind, Placebo-Controlled, Concentration-Escalating, Pharmacokinetic Study Evaluating the Systemic Absorption, Safety, and Efficacy of OMS201 in Subjects Undergoing Ureteroscopic Treatment of Ureteral- or Renal Collecting System-Located Stones
Brief Title: Pharmacokinetic, Safety and Efficacy Study of OMS201 in Subjects Undergoing Retrograde Ureteroscopic Removal of Upper Urinary Tract Stones
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C08-001
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Urinary Calculi; Urinary Stones; Urinary Tract Stones; Renal Calculi; Kidney Stones
Keywords: Urinary Calculi; Urinary Stones; Urinary Tract Stones; Renal Calculi; Kidney Stones; Calculi; Urolithotomy; Ureteroscopy
MeSH Terms: conditions — Urinary Calculi; Kidney Calculi; Calculi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Drug
  Interventions: Drug: OMS201
- 2 (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: OMS201 — Stage 1: OMS201 irrigation solution at 3X the base concentration during surgery
  Stage 2: OMS201 irrigation solution up to 10X the base concentration during surgery
  Arms: 1
Drug: Vehicle — Stages 1-2: Vehicle irrigation solution during surgery
  Arms: 2

SUMMARY:
The objectives of the study are to assess the systemic exposure, safety and efficacy of three concentrations of OMS201 in subjects undergoing retrograde ureteroscopic removal of upper urinary tract stones.

DETAILED DESCRIPTION:
The main objective is to estimate the systemic exposure of OMS201 in retrograde ureteroscopic treatment of upper urinary tract stones. Safety will be assessed by vital signs, laboratory values and adverse events. Exploratory efficacy measures will assess the effect of OMS201 on postoperative pain, duration of surgery and ease of placement of a ureteral access sheath.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years of age.
* Subject is undergoing retrograde ureteroscopic removal of renal-collecting system or ureteral stones for which general anesthesia will be used.

Exclusion Criteria:

* No allergies to any of the individual ingredients in OMS201.
* Subject taking a prohibited medication.
* Pregnant woman, nursing mother, or woman of child-bearing age unwilling to take contraception for the duration of the study.
* Subject who has had a renal transplant, has a single kidney, has compromised renal function, or has evidence of papillary necrosis.
* Subject who has evidence of a clinically significant urinary tract infection.
* Subject who has a prior history of open or laparoscopic urinary tract surgery, or a history of a ureteral stricture.
* Subject who has congenital anomalies that would engender an increased procedural safety risk.
* Subject with a history of clinically significant chronic or episodic hypotension.
* Subject's physical examination is significantly abnormal for purposes of the study as determined by the Investigator.
* Subject's screening laboratory evaluations are not within normal limits AND abnormal results are determined by the Investigator to be clinically significant.
* Subject is at risk from anesthesia.
* Subject is on chronic diuretic use.
* Subject has a present condition or history of any clinically significant medical disorder and is determined by the Investigator to be an unsuitable candidate for receipt of an investigational drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Peak systemic exposure. | Day of surgery

SECONDARY OUTCOMES:
Safety | Day 7
Degree of pain | 7 days
Duration of the operation | Day of surgery
Ease of placement of the ureteral access sheath | Day of surgery

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California Irvine Medical Center, Orange, California
  - Urology Center of Colorado, Denver, Colorado
  - Urology Associates, Nasville, Tennessee
  - Urology San Antonio Research, San Antonio, Texas